CLINICAL TRIAL: NCT03149757
Title: Connecting Youth and Young Adults to Optimize ART Adherence: Testing the Efficacy of the Youth Thrive Intervention
Brief Title: Connecting Youth and Young Adults to Optimize ART Adherence: YouTHrive Efficacy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of North Carolina (Other); University of Michigan (Other); Emory University (Other); Children's Hospital of Philadelphia (Other); Baylor College of Medicine (Other); Cook County Hospital (Other); Montefiore Medical Center (Other); University of South Florida (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-3136; 1U19HD089881 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections
Keywords: Treatment Adherence; Alcohol or Drugs; Behavioral; Internet; Adolescents; Young Adults; Social Support
MeSH Terms: conditions — HIV Infections; Treatment Adherence and Compliance; Behavior

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YouTHrive (Experimental): YouTHrive is a five-month technology-based intervention that uses peer-to-peer interaction, daily self-monitoring, and tailored content to address barriers to HIV medication adherence.
  Interventions: Behavioral: YouTHrive
- Thrive Tips (Active Comparator): Participants randomized to the control condition will receive a weekly email with static informational content about living with HIV and general well being.
  Interventions: Behavioral: Information-only Control

INTERVENTIONS:
Behavioral: YouTHrive — The YT website is a mobile-enhanced private social networking website. Participants on the site are anonymous and choose alternate usernames and personalized profile features for a new online identity within YT. The investigators designed YouTHrive to encourage social support, reduce isolation, improve HIV medication adherence, and promote general well being. The study involves rolling recruitment so that new members are continuously entering the intervention. Participants use YT for five months before "graduating" from the program. The core components of YT are: 1) peer-to-peer interaction in a shared feed; 2) daily monitoring of HIV medication adherence and real-time mood; 3) daily mixed-media content with strategies to improve medication adherence' and 4) goal setting and monitoring.
  Other Names: YT
  Arms: YouTHrive
Behavioral: Information-only Control — Participants will receive 21 emails, once per week, for five months. The emails will include static informational content relatable to YLWH, but informational content will not be focused on ART medication adherence.
  Arms: Thrive Tips

SUMMARY:
YouTHrive (YT) is a two-arm randomized control trial (RCT) to test the efficacy of an adapted version of the Thrive With Me (TWM) intervention for youth living with HIV (YLWH). In the RCT, intervention participants will have access to the full YouTHrive (YT) website- a mobile-enhanced private social networking website aimed at improving medication adherence for YLWH. The investigators will enroll up to 60 YLWH for formative work on YT, and 300 YLWH (15-24 years old) of all genders living in eight cities and randomize them to either the intervention condition or control condition. Assessments will be collected at baseline and 5-month follow-up.

DETAILED DESCRIPTION:
Youth between the ages of 13 and 24 accounted for 22% of all new HIV infections in 2015. Less than half (44%) of youth living with HIV (YLWH) in the US are estimated to be virally suppressed, which is a well recognized critical factor in individual health and non-infectiousness. Given the high demands of social identity development during adolescence and early adulthood, as well as the increasing use of social media as important and influential communication channels, there is an ongoing need for innovative programs that leverage current communication channels to foster social support for ART adherence behaviors.

The investigators developed a program first called Thrive With Me (TWM) as an intervention that leverages enhanced peer-to-peer interaction, ART adherence reminders and self-monitoring, and ART and HIV informational content to improve ART adherence. Given youth's broad acceptance and adoption of many of the components of the TWM intervention, and the critical need for novel and scalable ART adherence interventions for this population, we have adapted TWM for a younger audience and all genders in a program called YouTHrive (YT).

Focus groups will provide insights into what features and functions of the current TWM study youth like and dislike to assist intervention adaptation. The investigators will conduct focus groups in three cities (Houston, Bronx, and Chicago) and will recruit up to 16 YLWH per city, and use the results to develop the YT intervention. Ahead of the RCT, the investigators will conduct usability testing on YT to gain feedback about the developed intervention. The investigators will recruit 12 YLWH in six cities to use the intervention for a two-week period for usability testing.

The randomized controlled efficacy trial will compare YT (N=150) to a control group (N=150). YLWH in the control arm will receive weekly static information-only emails, compared to daily use of the dynamic YT social network site for the intervention group. Participants will be recruited from eight cities: Atlanta, New York, Chapel Hill, Charlotte, Chicago, Houston, Philadelphia, and Tampa. Assessments will be collected at baseline and 5-month follow-up.

Specific Aims include:

Primary Objective: In a 2-arm RCT (n=300), assess the efficacy of YouTHrive(YT) to promote higher treatment success at month 5 among YLWH, compared to an HIV information-only control condition, as defined by higher self-reported ART adherence (primary), higher percent suppressed viral load (secondary), and higher HIV care attendance (secondary).

H1: Participants in the YT intervention arm than in the information-only control arm will report higher ART adherence at the 5-month follow-up time point.

H2: A higher proportion of participants in the YT intervention arm than in the information-only control arm will have suppressed viral load at the 5-month follow-up time point.

H3: Participants in the YT intervention arm than in the information-only control arm will report higher HIV care attendance at the 5-month follow-up time point.

H4: A higher proportion of participants in the YT intervention arm than in the information-only control arm will demonstrate treatment success on a composite variable of primary and secondary outcomes.

Secondary Objective 1: Assess whether YT has more HIV treatment benefits for substance-using than non-substance-using YLWH.

H5: Among YLWH in the YT intervention arm, a higher proportion of substance-using participants will demonstrate improvement on primary and secondary outcomes, and a composite variable of these outcomes, at the 5-month follow-up time point compared to non-substance-using participants.

Secondary Objective 2: Examine whether YT has positive impacts on mental health and social support.

H6: Participants in the YT intervention arm will report lower depression and anxiety and higher social support at the 5-month follow-up time point compared to those in an information-only control arm.

ELIGIBILITY:
Inclusion Criteria:

1. 15-24 years of age at the enrollment visit;
2. HIV-positive status;
3. Residing in Chicago, Houston, NYC, Philadelphia, Atlanta, Tampa, or Raleigh/Durham/Chapel Hill areas and available to meet in-person or virtually with SRV staff for visits at baseline and 5-month follow-up assessment;
4. English-speaking (since the intervention will be in English);
5. Anticipated continuous internet access and SMS messaging for the intervention period (approximately 5 months);
6. Not enrolled in another ART adherence intervention research study at the time of screening;
7. Has or is willing to create an e-mail address to use during the study period;
8. Did not attend an iTech Youth Advisory Board (YAB) or Youth Advisory Council (YAC) meeting where the YouTHrive study was presented or YouTHrive study materials were discussed.

Exclusion Criteria:

1. Is younger than 15 years old or older than 24 years old at the enrollment visit;
2. does not have an HIV-positive status;
3. Does not reside in Chicago, Houston, NYC, Philadelphia, Atlanta, Tampa, or Raleigh/Durham/Chapel Hill areas and not available to meet with SRV staff for visits at baseline, and 5-month follow-up assessment;
4. Does not speak English;
5. Does not anticipate having continuous internet access and SMS messaging for the intervention period (approximately 5 months);
6. Is enrolled in another ART adherence intervention research study at the time of screening;
7. Does not have or is not willing to create an e-mail address to use during the study period;
8. Is a member of an iTech Youth Advisory Board (YAB) or Youth Advisory Council (YAC).

Participants who are or become pregnant during the study period will not be excluded.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, PhD, Study Chair — University of North Carolina; Patrick S Sullivan, PhD, Study Chair — Emory University; Keith J. Horvath, PhD, Principal Investigator — University of Minnesota; K. Rivet Amico, PhD, Principal Investigator — University of Michigan
Locations (7):
- United States (7):
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Cook County Hospital and Health Systems CORE Center, Chicago, Illinois
  - Montefiore Children's Hospital, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will assure the timely release and sharing of data two years after the publication of the main trial findings from the final dataset. Study variables will be available; however, the investigators will protect the rights and privacy of human subjects by redacting all identifiers from the data set. The de-identified data from this project will be available through individual requests directed to the Principal Investigator.

REFERENCES:
- [Derived] Horvath KJ, MacLehose RF, Martinka A, DeWitt J, Hightow-Weidman L, Sullivan P, Amico KR. Connecting Youth and Young Adults to Optimize Antiretroviral Therapy Adherence (YouTHrive): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jul 30;8(7):e11502. doi: 10.2196/11502. PMID 31364601

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | YouTHrive | Thrive Tips
Started | 103 | 105
Completed | 96 | 100
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | YouTHrive | Thrive Tips | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.97 (2.34) | 21.32 (2.21) | 21.15 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 50
  Male | 74 | 84 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 64 | 68 | 132
  White | 14 | 19 | 33
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) of Self-Reported Antiretroviral Adherence
Description: Participants were presented with a visual analog scale (VAS) of the percentage of antiretroviral therapy (ART) adherence in the past 30 days on a scale from 0% to 100% (with 10% increments as response options) and asked to choose the level of ART adherence they achieved in the past 30 days. The mean percentage of ART adherence across all participants was calculated.
Time Frame: 5-month follow-up
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | YouTHrive | Thrive Tips
Number analyzed (Participants) | 77 | 77
Unit on a scale | 85.71 (19.29) | 85.53 (16.4)

2. Secondary Outcome: Percentage of Participants With Undetectable HIV Viral Load
Description: HIV viral load was abstracted from participants' medical records or a blood draw as part of research protocols (if no recent viral load measure was available from the medical record). A participant was recorded as having an undetectable HIV viral load if the level of HIV was so low that the test used by that clinic did not detect HIV in the participant (between <20 and <50 HIV copies depending on the clinic's viral load test).
Time Frame: 5-month follow-up
Population: The number of participants on which the study team was able to collect HIV viral load measure on was lower than the number of participants who completed the self-report surveys. As such, the number reported on for HIV viral load is smaller than the number of participants available for the primary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | YouTHrive | Thrive Tips
Number analyzed (Participants) | 65 | 55
Participants | 56 | 43

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | YouTHrive | Thrive Tips
All-Cause Mortality (participants affected / at risk) | 1/103 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/105
Other Adverse Events (participants affected / at risk) | 0/103 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03149757/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03149757/ICF_001.pdf